CLINICAL TRIAL: NCT00552383
Title: The Impact of Developmental Care in the Neonatal Intensive Care Unit: The Edmonton Randomised Controlled Trial of NIDCAP (Newborn Individualised Developmental Care and Assessment Program)
Brief Title: The Edmonton Randomised Controlled Trial of NIDCAP - Based Developmental Care
Acronym: NIDCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Canadian Lung Association (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199700189 (AHFMR); 199700189 (AHFMR)
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Infant, Premature
Keywords: Preterm Infant; Behaviour; Developmental Care; NIDCAP; Family Centred Care; Neurodevelopmental Outcome, preterm infant
MeSH Terms: conditions — Premature Birth; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: NIDCAP based developmental care — Infants in the intervention arm will receive care in the NICU by nursing staff who have received basic education in NIDCAP - based developmental care. They will also have NIDCAP behavioural observations performed by NIDCAP - Certified staff [this includes 3 of the investigators], at intervals during their stay at the study site NICU. These behavioural observations form the basis for behaviourally guided "baby -friendly" care, so that the timing and pace of caregiving is synchronised to the infant's readiness. Parents are actively encouraged to become the infant's primary caregiver in the NICU.

SUMMARY:
NIDCAP based developmental care is a method of looking after preterm infants that is guided by the infant's behavioural cues, and that actively involves parents in the care of their infant. There is limited evidence that outcomes for infants are improved if they receive NIDCAP based care. This study evaluates the effects of introducing NIDCAP based care to a level III neonatal intensive care unit, in the post - surfactant era, and also evaluates its effects on developmental outcomes at age 18 months.

DETAILED DESCRIPTION:
This RCT differs from previous trials in that it is conducted in the post - surfactant era [an intervention that has greatly changed clinical neonatology]. The number of infants required to demonstrate a clinically relevant outcome [Length of Hospital Stay] has been calculated a priori. The infants will be tracked for outcome data after transfer to peripheral nurseries [a reality in today's healthcare environment], allowing generalisability of results to other high risk, referral Neonatal Intensive Care units. Neurodevelopmental outcomes will be evaluated at 18 months; [these data are sparse from previous studies]. This RCT will therefore demonstrate whether NIDCAP based care is truly an effective intervention for the very low birth weight infant.

ELIGIBILITY:
Inclusion Criteria:

* birth weight between 500g to <1250g
* gestational age </= 32 weeks
* birth weight between 3rd to 97th percentile for gestational age
* survival to >48 hr age
* at least one parent speaks English or a language spoken by study investigator
* twins eligible if BOTH meet all criteria

Exclusion Criteria:

* chromosomal abnormalities
* major congenital anomalies
* maternal drug and /or alcohol use in pregnancy
* congenital infection
* decision made to withdraw intensive care treatments, or discussion about this already initiated with family

Ages: 2 Days to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 1998-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Sept 1999 to Dec 2002

SECONDARY OUTCOMES:
Days of ventilation | Sept 1999 to Dec 2002
Incidence of Chronic Lung Disease of Prematurity | Sept 1999 to Dec 2002
Neurodevelopmental Disability at corrected age 18 months | April 2001 to Dec 2004
incidence of sepsis | Sept 1999 - Dec 2002
Use of sedative medication | sept 1999 - dec 2002
Maternal Stress | Sept 1999 - Dec 2002
incidence of Apnea of Prematurity | sept 1999 - dec 2002
time to regain birthweight | sept 1999 - dec 2002
time to attain full enteral feeds | sept 1999 - dec 2002
incidence of intracranial hemorrhage and periventricular leukomalacia | sept 1999 - dec 2002

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine L Peters, MN PhD, Principal Investigator — University of Alberta, Faculty of Nursing
Locations (1):
- Royal Alexandra Hospital, Neonatal Intensive Care Unit, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Als H, Lawhon G, Duffy FH, McAnulty GB, Gibes-Grossman R, Blickman JG. Individualized developmental care for the very low-birth-weight preterm infant. Medical and neurofunctional effects. JAMA. 1994 Sep 21;272(11):853-8. PMID 8078162
- [Background] Als H, Lawhon G, Brown E, Gibes R, Duffy FH, McAnulty G, Blickman JG. Individualized behavioral and environmental care for the very low birth weight preterm infant at high risk for bronchopulmonary dysplasia: neonatal intensive care unit and developmental outcome. Pediatrics. 1986 Dec;78(6):1123-32. PMID 3786036
- [Background] Westrup B, Kleberg A, von Eichwald K, Stjernqvist K, Lagercrantz H. A randomized, controlled trial to evaluate the effects of the newborn individualized developmental care and assessment program in a Swedish setting. Pediatrics. 2000 Jan;105(1 Pt 1):66-72. doi: 10.1542/peds.105.1.66. PMID 10617706
- [Background] Fleisher BE, VandenBerg K, Constantinou J, Heller C, Benitz WE, Johnson A, Rosenthal A, Stevenson DK. Individualized developmental care for very-low-birth-weight premature infants. Clin Pediatr (Phila). 1995 Oct;34(10):523-9. doi: 10.1177/000992289503401003. PMID 8591679
- See also: the NIDCAP education and training program is described; accredited NIDCAP training centres are listed here also — http://www.nidcap.com/